CLINICAL TRIAL: NCT03568695
Title: Detection of Chlamydia Trachomatis, Neisseria Gonorrhoeae and Mycoplasma Genitalium by Real-time Multiplex Polymerase Chain Reaction After Pooling Pharyngeal, Anorectal and Urinary Samples, in Men Who Have Sex With Men
Brief Title: Detection of Chlamydia Trachomatis, Neisseria Gonorrhoeae and Mycoplasma Genitalium by Real-time Multiplex Polymerase Chain Reaction (PCR) After Pooling Pharyngeal, Anorectal and Urinary Samples
Acronym: ISTPOOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2018-01
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Chlamydia Trachomatis Infection; Neisseria Gonorrheae Infection; Mycoplasma Genitalium Infection; Sensitivity; Polymerase Chain Reaction
Keywords: pooled analysis; sensitivity; men who have sex with men
MeSH Terms: conditions — Gonorrhea; Hypersensitivity; Homosexuality | interventions — Urination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Detected patients (Other): If they agree to participate in the study, the patients detected for one or the other of the STIs (Chlamydia trachomatis, Neisseria gonorrhoeae, Mycoplasma genitalium) on one site, will have on day of result return, two new samples on each of the three sites (pharynx, rectum, urine) which will make it possible to compare the difference of sensitivity between real-time multiplex PCR from pools of 3 samples and the usual technique .
  Interventions: Diagnostic Test: Two samples on each of the three sites (pharynx, rectum, urine)

INTERVENTIONS:
Diagnostic Test: Two samples on each of the three sites (pharynx, rectum, urine) — two new samples on each of the three sites (pharynx, rectum, urine) which will make it possible to compare the difference of sensitivity between real-time multiplex PCR from pools of 3 samples and the usual technique .

SUMMARY:
This study aims to compare the sensitivity of detecting Chlamydia trachomatis, Neisseria gonorrhoeae and Mycoplasma genitalium by real-time multiplex PCR in a pooled analysis (i.e. gathering pharyngeal, anorectal and urinary samples) versus the standard of care (where a real-time multiplex PCR is made in each of the three samples).

DETAILED DESCRIPTION:
Patients detected positive for one of the three (Sexually Transmitted Infection)STIs (Chlamydia trachomatis, Neisseria gonorrhoeae or Mycoplasma genitalium) on one site will be re-sampled twice at each of the three sites (pharynx, rectum, urine) before receiving antibiotics. Then, a real-time multiplex PCR will be performed on the pooled sample (merging pharyngeal, anorectal and urinary samples) versus on each of the three samples separately (i.e. standard of care) to compare both sensitivities.

ELIGIBILITY:
Inclusion Criteria:

* Patient having provided a written consent;
* Patient age > 18 years;
* Man who have sex with men tested positive for one the three STIs : Chlamydia trachomatis, Neisseria gonorrhoeae or Mycoplasma genitalium
* Covered by health insurance

Exclusion Criteria:

* Being under tutorship
* Being deprived of liberty
* Patient who received antibiotic treatment prior to study inclusion and re-sampling

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
To evaluate the sensitivity of Chlamydia trachomatis, Neisseria gonorrhoeae and Mycoplasma genitalium detection in a pooled analysis | Day 1
  Sensitivity rates will be compared using non parametric statistical analysis. The pooling method will be considered as acceptable if the sensitivity reach at least 95%.

SECONDARY OUTCOMES:
Impact of the strategies on the costs | Day 1
  Costs will include time of lab staff, DNA extraction, PCR material in the two strategies and related to 1000 patients

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PRAZUCK, Dr, Principal Investigator — CHR d'Orléans
Locations (5):
- France (5):
  - CH de Niort, Niort
  - CHR d'Orleans, Orléans
  - CHU de Poitiers, Poitiers
  - CH Laennec, Quimper
  - CHU de Tours, Tours

REFERENCES:
- [Background] Kacena KA, Quinn SB, Howell MR, Madico GE, Quinn TC, Gaydos CA. Pooling urine samples for ligase chain reaction screening for genital Chlamydia trachomatis infection in asymptomatic women. J Clin Microbiol. 1998 Feb;36(2):481-5. doi: 10.1128/JCM.36.2.481-485.1998. PMID 9466763
- [Background] La Ruche G, Le Strat Y, Fromage M, Bercot B, Goubard A, de Barbeyrac B, Sednaoui P, Cambau E, Lot F. Incidence of gonococcal and chlamydial infections and coverage of two laboratory surveillance networks, France, 2012. Euro Surveill. 2015 Aug 13;20(32):6-15. PMID 26290487
- [Background] Lewis JL, Lockary VM, Kobic S. Cost savings and increased efficiency using a stratified specimen pooling strategy for Chlamydia trachomatis and Neisseria gonorrhoeae. Sex Transm Dis. 2012 Jan;39(1):46-8. doi: 10.1097/OLQ.0b013e318231cd4a. PMID 22183846
- [Background] Kacena KA, Quinn SB, Hartman SC, Quinn TC, Gaydos CA. Pooling of urine samples for screening for Neisseria gonorrhoeae by ligase chain reaction: accuracy and application. J Clin Microbiol. 1998 Dec;36(12):3624-8. doi: 10.1128/JCM.36.12.3624-3628.1998. PMID 9817885
- [Derived] Prazuck T, Lanotte P, Le Moal G, Hocqueloux L, Sunder S, Catroux M, Garcia M, Perfezou P, Gras G, Plouzeau C, Leveque N, Beby-Defaux A. Pooling Rectal, Pharyngeal, and Urine Samples to Detect Neisseria gonorrhoeae, Chlamydia trachomatis, and Mycoplasma genitalium Using Multiplex Polymerase Chain Reaction Is as Effective as Single-Site Testing for Men Who Have Sex With Men. Open Forum Infect Dis. 2022 Oct 31;9(10):ofac496. doi: 10.1093/ofid/ofac496. eCollection 2022 Oct. PMID 36324326